CLINICAL TRIAL: NCT01020591
Title: The Effect of Osteopathic Manual Therapy on the Vascular Supply to the Lower Extremity in Individuals With Knee Osteoarthritis, a Randomized Trial
Brief Title: The Effect of Osteopathic Manual Therapy on Vascular Supply
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Wendy Jardine, Physiotherapist osteopath, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA-RS/2010-227
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; manual therapy; osteopathy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic evaluation (Active Comparator): osteopathic evaluation of motion and tissue mobility
  Interventions: Other: Osteopathic evaluation
- Osteopathic evaluation with treatment (Experimental): osteopathic evaluation of motion and tissue mobility followed by osteopathic manual therapy release of the tight or restricted tissues
  Interventions: Other: Osteopathic evaluation with treatment

INTERVENTIONS:
Other: Osteopathic evaluation — evaluation of movement and tissue mobility
  Arms: Osteopathic evaluation
Other: Osteopathic evaluation with treatment — osteopathic evaluation followed by osteopathic manual therapy release of tissues identified as tight or restricted
  Arms: Osteopathic evaluation with treatment

SUMMARY:
The purpose of this study is to determine if the use of osteopathic manual therapy can influence the vascular supply to the knee, knee range of motion, balance and knee pain, in a group of subjects with knee osteoarthritis. It is also the objective of this study to determine if there is a difference between the osteopathic evaluation and the combination of an osteopathic evaluation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic-confirmed knee osteoarthritis

Exclusion Criteria:

* Subjects who are unable to ambulate independently (without an aid) and safely the distance of a city block
* Subjects who have an uncontrolled medical condition (e.g. heart (angina) or respiratory condition (asthma))
* Subjects who have a neurological condition (e.g. Parkinson's, Multiple Sclerosis)
* Subjects who have both knees affected by osteoarthritis and have had previous surgery to both knees
* Subjects who have knee OA in only one knee and that knee has had previous knee surgery
* Subjects who have previous vascular surgery to either leg

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Jardine, MScPT, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty subjects between the age of 48 and 80 years with radiographic confirmed knee OA were recruited. All data collection took place at the School of Health Sciences Room 658 Bethune building on South park St in Halifax Nova Scotia between January and March of 2010.
Groups:
- Osteopathic Evaluation: osteopathic evaluation: forward flexion test, hip drop test, the sitting forward flexion test, sitting diaphragm evaluation, sphenobasilar symphysis (SBS) listening, sacral listening, pelvic floor evaluation, peritoneal bag evaluation and global femoral artery evaluation
Period: Overall Study
Arm/Group | Osteopathic Evaluation | Osteopathic Evaluation With Treatment
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osteopathic Evaluation | Osteopathic Evaluation With Treatment | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.73 (9.63) | 63.20 (7.97) | 63.47 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Resistive Index (RI)
Description: Ultrasonographic examination provides a non-invasive method to assess blood flow dynamics. The resistive index (RI), calculated from arterial blood flow velocities, reflects vascular resistance. The RI was calculated by dividing the peak systolic velocity (PSV) minus the end-diastolic velocity by the peak systolic velocity, and is cited frequently in the literature for measuring hemodynamics of peripheral vessels.
Time Frame: Participants attended one visit; The outcome measure (RI) was before and after an osteopathic session on the same day; The data collection of the 30 subjects took place between Jan to March 2010; each subject had outcomes measured on one day
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Pre Test to the Osteopathic Evaluation; Same Day Post Test to Osteopathic Evaluation: osteopathic evaluation: forward flexion test, hip drop test, the sitting forward flexion test, sitting diaphragm evaluation, sphenobasilar symphysis (SBS) listening, sacral listening, pelvic floor evaluation, peritoneal bag evaluation and global femoral artery evaluation
- Pre Test to the Osteopathic Evaluation With Treatment; Post Test to Osteopathic Evaluation With Treatment: osteopathic evaluation of motion and tissue mobility followed by osteopathic manual therapy release of the tight or restricted tissues
Arm/Group | Pre Test to the Osteopathic Evaluation | Pre Test to the Osteopathic Evaluation With Treatment | Same Day Post Test to Osteopathic Evaluation | Post Test to Osteopathic Evaluation With Treatment
Number analyzed (Participants) | 15 | 15 | 15 | 15
ratio | 1.30 (0.07) | 1.40 (0.09) | 1.30 (0.06) | 1.35 (0.08)
Statistical Analysis 1: Comparison: Pre Test to the Osteopathic Evaluation vs Pre Test to the Osteopathic Evaluation With Treatment vs Same Day Post Test to Osteopathic Evaluation vs Post Test to Osteopathic Evaluation With Treatment; A two factor mixed model Analysis of Variance (ANOVA) for Group (Evaluation vs. Treatment) with repeated measures (pre vs. post test) was employed to test for main effects and all interactions for the Resistive Index; Test type: Non-Inferiority or Equivalence — The power and sample size calculations, based on the ability to detect treatment and evaluation group differences, were performed on Minitab™ V.15. 40 participants were estimated to be required for group allocation (20 in each group: evaluation;evaluation and treatment)for 80% power in at least 3 out of the 4 outcome measures. After 30 subjects, analysis determined that there would be no further statistically significant changes in results therefore, data collection was stopped at 30 subjects; p < 0.05, ANOVA

2. Secondary Outcome: The Knee Flexion Active Range of Motion, Balance and Pain (VAS)
Time Frame: Jan 2010 to March 2010
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Jan 2010 to March 2010
Arm/Group | Osteopathic Evaluation | Osteopathic Evaluation With Treatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No